CLINICAL TRIAL: NCT06569719
Title: Effectiveness of Complex Decongestive Therapy for the Treatment of Lymphedema in Breast Cancer Patients Who Received Lymphovenous Anastomosis Surgery: a Pilot Study
Brief Title: Effectiveness of CDT for the Treatment of Lymphedema in Breast Cancer Patients Who Received LVA Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Universitaria Maria Cano (Other)
Responsible Party: Principal Investigator, Catalina Lopera Muñetón, Clinical professor, Advanced Bionics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 013008013-2023-311
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients who have recieved lymphovenous anastomosis in the past 12 months and participates in complex decongestive therapy (CDT), including all its techniques, consisting of a total of 10 therapy sessions and a follow-up at 3 months
  Interventions: Other: Complex decongestive therapy
- Control (No Intervention): Patients received lymphovenous anastomosis and they are provided with compression garments as part of the treatment withot recieving CDT . This group will have an initial assessment and follow-up at 3 months

INTERVENTIONS:
Other: Complex decongestive therapy — Includes manual lymphatic drainage (MLD), compression therapy (which consists of compression bandages, compression sleeves, or other types of compression garments), skin care, and lymph-reducing exercises
  Arms: Intervention

SUMMARY:
Breast cancer is the most common type of cancer in women worldwide. Advances in treatment have increased survival rates, so patients must live with the complications resulting from the cancer and its treatment. One of the most common side effects is lymphedema, which can occur as a secondary effect of surgical or radiotherapy treatment. Lymphatic edema is a condition characterized by an excess of lymphatic fluid, rich in proteins, in the subcutaneous tissue, causing pain, a feeling of heaviness in the affected limb, restricted range of motion, and, in some cases, progressing to the formation of ulcers and recurrent infections; inevitably affecting the quality of life of the women who suffer from it. There are various therapeutic strategies to reduce the risk of developing lymphedema or to treat it. Among the management options is complex decongestive therapy (CDT), which is a conservative treatment that includes manual lymphatic drainage (MLD), compression therapy, skin care, and lymph-reducing exercises (LRE). Surgical options include lymph node transfer and lymphovenous anastomosis; redirecting lymphatic circulation and reducing edema in the affected limb. This is why the current research is undertaken, aiming to evaluate the effectiveness of combining these two treatment approaches in terms of reducing lymphedema, the presence of cellulitis, and changes in patients' quality of life

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer among women, with an estimated 2.3 million new cases diagnosed worldwide in 2020, with especially high incidence in developed countries. The five-year survival rate for breast cancer exceeds 90%, and the average ten-year survival rate for women with non-metastatic invasive breast cancer is 84% (Ferlay et al., 2021).

As a consequence, there is an increasing number of women facing early and late side effects from breast cancer treatment. One of the most common side effects is lymphedema, with a reported incidence after cancer treatment around 30% (Martínez Jaimez, 2017). In Colombia, it is estimated that 28% of women who undergo lymphadenectomy develop lymphedema (Valencia Legarda et al., 2020). Lymphedema is a chronic inflammatory disease that affects approximately 250 million people worldwide, mostly associated with cancer treatment. It can occur as a result of breast cancer surgery and/or radiotherapy (Riady-Aleuy et al., 2022). Lymphedema is defined as the accumulation of protein-rich fluid in the interstitium, secondary to abnormalities in the lymphatic transport system.

According to the impact of lymphedema on the quality of life of individuals, as well as the associated social and economic costs, efforts must be made to prevent and treat it. Various conservative strategies are used to reduce the risk of developing lymphedema and to manage it once it has developed. Among the physiotherapeutic options is complex decongestive therapy (CDT), which is a conservative treatment that includes manual lymphatic drainage (MLD), compression therapy (consisting of compression bandages, compression sleeves, or other types of compression garments), skin care, and lymph-reducing exercises (LRE).

Another treatment option is surgery, which has traditionally been considered a last resort when conservative measures have failed. However, increasingly advanced surgical interventions are now being performed early in the disease process, with the hope of preventing or reversing edema that arises from impaired lymphatic flow (Markkula et al., 2019). These interventions include liposuction, lymph node transfer, and lymphaticovenular anastomosis (LVA). The latter was first described in 1960, but it wasn't until 1989 in Japan and in 2020 in Colombia that it became the gold standard of microsurgery, emerging as an innovative technique in our field, increasingly used as a treatment for lymphedema rather than as a last-resort strategy when other treatments have failed (Gupta et al., 2021).

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphedema due to cancer.
* Patients who have undergone lymphovenous anastomosis surgery in the past 12 months

Exclusion Criteria:

* Decompensated heart failure
* Decompensated renal failure
* Open wounds
* Decompensated arterial insufficiencies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Lymphedema change | Baseline, post-intervention up to 3 weeks and 3 months follow up
  Upper and leg Extremity Lymphedema Index. The index includes 5 perimeters that are sum and divided by BMI. Classified as mild leg lymphedema < 250, mild to severe 250-350 and severe > 350. Classified as mild arm lymphedema < 130, mild to severe 130-150 and severe > 150 This outcome is compound by multiple measurements that will be aggregated to arrive at one reported.

SECONDARY OUTCOMES:
Quality of life change | Baseline, post-intervention up to 3 weeks and 3 months follow up
  ARM and LEG Lymphoedema Quality of Life Tool (LYMQOL). It includes 3 domains (Function, symptoms, mood) and an overall quality of life score. Domain totals are calculated by adding the individual scores and dividing the total by the number of questions answered. A higher number means a poor quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Fundación Universitaria María Cano, Medellín, Antioquia
  - Fundación Universitaria María cano, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in cancer lymphedema. Data or samples shared will be coded. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will made accessible for up to 18 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact catalinaloperamuneton@fumc.edu.co